CLINICAL TRIAL: NCT02834208
Title: Neurofunctional Basis of Emotion Processing: Clinical, Genetic, Biological and Imaging Study in Patients With Schizophrenia and Healthy Relatives of Patients in Comparison With a Control Group
Brief Title: Emotion Endophenotypes in Schizophrenia
Acronym: SCHIZOIMAGEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-38; 2015-A01475-44 (Other: ANSM)
Record Dates: First submitted 2016-07-04; First posted 2016-07-15 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Magnetic Resonance Spectroscopy; Polymorphism, Genetic; Polymorphism, Single Nucleotide; DNA; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Schizophrenia subjects (Experimental): 35 patients suffering from schizophrenia
  Interventions: Other: MRI (Magnetic resonance imaging); Genetic: Polymorphism (SNP in DNA); Genetic: quantitative measures of mRNA; Other: Neuropsychological assessment
- Healthy siblings (Other): 35 healthy siblings of the patients suffering from schizophrenia
  Interventions: Other: MRI (Magnetic resonance imaging); Genetic: Polymorphism (SNP in DNA); Genetic: quantitative measures of mRNA; Other: Neuropsychological assessment
- Healthy controls (Other): 35 healthy "controls "patients
  Interventions: Other: MRI (Magnetic resonance imaging); Genetic: Polymorphism (SNP in DNA); Genetic: quantitative measures of mRNA; Other: Neuropsychological assessment

INTERVENTIONS:
Other: MRI (Magnetic resonance imaging)
Genetic: Polymorphism (SNP in DNA)
Genetic: quantitative measures of mRNA
Other: Neuropsychological assessment

SUMMARY:
Schizophrenia is an invalidating psychiatric illness with a strong genetic component characterized by abnormal processing of emotional information. This alteration in emotion processing has been described in acute as well as in remission phases of the illness. It has also been found in healthy relatives of patients with schizophrenia and in subjects at high risk of psychosis. Thus, alterations in emotional information processing are not only linked to the prognosis but can also be considered as a marker of vulnerability of schizophrenia. In addition, schizophrenia patients differ from healthy controls in neural activity in brain regions implicated in emotions processing. However, interpretation of findings in patients is limited by confounding factors, such as antipsychotic treatments or alterations due to the course of illness. Also, there is no data concerning genetic factors (polymorphisms or gene expression) underlying these patterns of cerebral activation in emotion information processing.

So, the main objective of this study is to compare the cerebral activity of schizophrenia patients to that of healthy siblings and healthy controls in an emotional processing task.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant, right-handed, aged from 18 to 45 years old
* Haven given their written consent
* DSM-5 (Diagnostic and Statistical Manual of Mental Disorders version 5) diagnosis of schizophrenia
* Remitted phase (criteria of Andreasen)
* Stable doses of antipsychotics during the last 6 weeks
* No severe somatic illness
* Normal clinical exam
* Inscription to the social security

Exclusion Criteria:

* Women in genitally active period without contraception
* Women pregnant or breast feeding
* Participants presenting a severe somatic /neurologic condition
* Present/history in the last year of alcohol or drug abuse
* Participating in another clinical study or still in period of exclusion of a previous clinical trial
* Contraindication to an MRI test (metallic foreign body, pacemaker, heart valve, chirurgical clip, claustrophobia…)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygen Level dependent (BOLD) signal activity in Anterior Cingulate Cortex (ACC) measured by functional MRI | 4 hours

SECONDARY OUTCOMES:
Assessment of the functional connectivity in cortico-limbic circuit which underlie the emotional information using functional MRI | 4 hours
Description of whole brain neuro-anatomy based using Voxel Brain Morphometry (VBM) | 4 hours
Quantitative expression of messenger Ribo Nucleic Acid (mRNA) in Peripheral Blood Mononuclear Cells (PBMC) | 4 hours
Polymorphism (single-nucleotide polymorphism SNP) of DNA (DeoxyriboNucleic Acid) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Pôle Psychiatrie Centre CHU Conception, Marseille, APHM, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided